CLINICAL TRIAL: NCT05618145
Title: Multicenter, Nationwide, Observational, Prospective Study Based on the Development of a Primary Sclerosing Cholangitis Patient's Database Linked to a Biological Sample Storage
Brief Title: National Database on Primary Sclerosing Cholangitis (PSC)
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: PSC_Database
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary Sclerosing Cholangitis; Disease phenotypes; National Database
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples are collected at time of recruitment (blood, urine and liver tissue).The collection of liver tissue depends on the specific procedures that are performed based on clinical needs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PSC population residing in Italy: All PSC patients living in Italy and aged at least 17 years can be included in the database.
  Interventions: Other: Clinical information

INTERVENTIONS:
Other: Clinical information — The investigators will recruit PSC patients and collect important clinical information and laboratory investigation, together with biological samples.

SUMMARY:
Primary sclerosing cholangitis (PSC) a rare, chronic fibroinflammatory disease of the liver.

No data about the disease epidemiology exist in Italy. Therefore this study aims to develop a national PSC patient database linked to a biological sample storage.

DETAILED DESCRIPTION:
Primary sclerosing cholangitis is a chronic fibroinflammatory disease of the liver characterized by chronic inflammation and sclerosis of the intrahepatic and/or extrahepatic bile ducts, and a risk for progression to liver failure and development of colorectal and hepatobiliary cancer 1. Both children and adults are affected. Patients with PSC have a diminished life expectancy with a median survival of 17 years after diagnosis. PSC is the leading indication for transplantation in some European countries. Epidemiological studies have found the highest prevalence rates of PSC in Northern European countries and North America (United States and Canada) ranging between 3.85 to 16.2 per 100,000 persons. In Italy, the estimates is of 0.8 per 100,000 persons but these figures underestimate the real disease burden 2.

Liver transplantation is currently the only life-extending accepted therapy for patients with end-stage liver disease (ESLD) secondary to PSC, and patients with PSC complicated by CCA who meet specific criteria. PSC recurs in the transplanted liver in up to 40% of patients. Taken together and combined with patients' debilitating quality of life issues, these data highlight the considerable disease burden and clinical impact of PSC on patients' outcomes. There is a strong, yet poorly understood, relationship between PSC and IBD; nearly 70%-80% of PSC patients have IBD, mainly ulcerative colitis.

Despite the high mortality associated with PSC and the efforts to optimize its management, there is no medical therapy proven to halt the progression of PSC or prevent its serious complications.

There have been no epidemiologic studies in PSC carried out in Italy, with the exception of the report of prevalence from the National registry of rare disease which provided an underestimated prevalence of 500 patients across the country. However, this study is limited by the nature of the registry which has administrative purposes and has a high rate of underreported cases.

The aim of the study is to implement a nationwide data collection on this rare disease to describe incidence and prevalence of PSC in Italy; identify and define distinct phenotypes and sub-phenotypes of PSC patients; identify factors influencing the progression of PSC and affecting mortality; assess safety and long-term efficacy of novel therapies.

The investigators will recruit patients and organise the collection of important clinical information and laboratory investigation, together with biological samples. Data will be collected in the form of electronic Case Report Forms (REDCap cloud) that will be completed by clinicians at baseline and thereafter on an annual basis. The clinical information will allow us to identify patients' clinical profiles. The biological samples will allow to understand key aspects of people's make up.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent prior to any study specific procedure being performed;
* Diagnosis of PSC according to the most recent published guidelines (EASL);

Exclusion Criteria:

* Subject unwilling to participate at the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All PSC patients living in Italy and aged at least 17 years can be included in the database. Willing and able to give informed consent prior to any study specific procedure being performed; Diagnosis of PSC according to the most recent published guidelines (EASL).
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2032-10-21 (Estimated); Study Completion 2032-10-21 (Estimated)

PRIMARY OUTCOMES:
Identify and define distinct phenotypes and sub-phenotypes of PSC patients at higher risk of disease progression. | Overall duration of the study (10 years)
  Identify and define distinct phenotypes and sub-phenotypes of PSC patients at higher risk of disease progression.

SECONDARY OUTCOMES:
Identification of factors associated with response to therapies; | Overall duration of the study (10 years)
  Identification of factors associated with response to therapies;
Identification of biomarkers influencing the progression of PSC and affecting mortality | Overall duration of the study (10 years)
  Identification of biomarkers influencing the progression of PSC and affecting mortality
Assessment of safety and long-term efficacy of novel therapies | Overall duration of the study (10 years)
  Assessment of safety and long-term efficacy of novel therapies

CONTACTS AND LOCATIONS:
Locations (63):
- Italy (63):
  - Ospedali riuniti di Ancona, Ancona
  - Policlinico di Bari, Bari
  - ASST Bergamo ovest, Bergamo
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale Sant'Orsola Malpighi, Bologna
  - Policlinico S. Orsola Malpighi, Bologna
  - Azienda sanitaria dell'Alto Adige, Bolzano
  - Spedali civili, Brescia
  - Unità epatologica ed ecografia internistica a valenza dipartimentale, Fondazione Ospedaliera Poliambulanza, Brescia
  - Policlinico universitario Monserrato, Cagliari
  - Presidio Ospedaliero San Michele ARNAS G. Brotzu, Cagliari
  - Osp. "S de Bellis" - IRCCS, Castellana Grotte
  - UO epatologia Ospedale Garibaldi, Catania
  - Azienda Ospedaliera Universitaria Mater Domini, Catanzaro
  - Azienda Ospedaliera Universitaria- Mater Domini, Catanzaro
  - Ospedale Valduce, Como
  - Unità operativa complessa di medicina interna- Azienda ospedaliera di Cosenza, Cosenza
  - ASST di Cremona, Cremona
  - Ospedale santa croce, Cuneo
  - Presidio Ospedaliero di Faenza (RA), Faenza
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Azienda ospedaliera universitaria careggi Firenze, Florence
  - Azienda ospedaliera universitaria Careggi, Florence
  - Centro C.U.R.E. Centro Universitario per la ricerca e la Cura delle Malattie Epatiche, Foggia
  - Ospedale Casa Sollievo della Sofferenza, Foggia
  - ASST Valle Olona, Gallarate
  - Policlinico San Martino, Genova
  - Presìdio Ospedaliero "Giovanni Paolo II", Lamezia Terme
  - ASST Lecco, Lecco
  - UO di epatologia clinica e biomolecolare. Università degli studi di Messina, Messina
  - Az. Ospedaliera San Paolo- Polo universitario, Milan
  - Istituto scientifico universitario San Raffaele, Milan
  - Ospedale Niguarda Ca' Granda, Milan
  - Ospedale San Giuseppe, Milan
  - Policlinico di Milano, Milan
  - Dipartimento Ospedaliero di Medicina Interna, Modena
  - ASST Monza, Monza
  - Fondazione Evangelica Villa Betania, Ospedale generale di Zona, Napoli
  - Ospedale policlinico Federico II di Napoli, Napoli
  - Università della Campania Luigi Vanvitelli, Napoli
  - Ospedale maggiore della carità, Novara
  - Azienda Ospedaliera di Padova, Padua
  - UO di Gastroenterologia Azienda ospedaliera di Padova, Padua
  - Policlinico Paolo Giaccone, Palermo
  - Azienda ospedaliero universitaria di Parma, Parma
  - Istituto Clinico Città di Pavia-Gruppo Sandonato, Pavia
  - Azienda ospedaliera di Perugia, Perugia
  - Day Hospital Internistico e ambulatorio di Epatologia, ASL Pescara, Pescara
  - Aou pisana Cisanello, Pisa
  - Ospedale di Pordenone AS FO, Pordenone
  - Ospedale San Carlo, Potenza
  - Azienda unità sanitaria locale della Romagna, Rimini
  - Ospedale A. Gemelli, Roma
  - Policlinico Umberto I, Roma
  - Policlinico universitario campus bio-medico, Roma
  - Universita' di Roma Tor Vergata, Roma
  - Istituto clinico Humanitas, Rozzano
  - Università degli studi di Salerno, Salerno
  - Azienda Ospedaliero-Universitaria Molinette, Torino
  - Azienda provinciale per i servizi sanitari, Trento
  - Ospedale di Cattinara, ASU GI, Trieste
  - ASU FC, Udine
  - ASST Sette Laghi, Varese